CLINICAL TRIAL: NCT03583749
Title: Pharmacokinetics and Safety of Antimicrobial Agents Administered by Subcutaneous Route in Patients AGEd Over 65 Years
Acronym: PhASAge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2017/37
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Antimicrobials; Subcutaneous Injection; Antibiotic; Older People
Keywords: Antimicrobial agents; subcutaneous administration; safety; pharmacokinetics; elderly
MeSH Terms: interventions — Injections, Subcutaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The sampling times chosen are the following:
  * C0: concentration measured at the end of the therapeutic interval, just before the following infusion, which corresponds to the minimum or residual concentration
  * Cperf: concentration measured at the end of infusion: immediately after stopping the infusion, which corresponds to the maximum concentration IV
  * C5h: concentration measured in the elimination phase, 5h after the end of the infusion. For the subcutaneous route only, an additional sample will be taken:
  * C2h: concentration measured 2h after the end of the SC infusion.
  The tubes will then be processed in the local pharmacokinetic laboratory as follows:
  For each antibiotic, the blood samples obtained from each recruitment center will be transported, centrifuged, aliquoted and frozen at the local pharmacology laboratory. The tubes will then be batched to the centralized transport dosing laboratory every 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- amoxicillin-clavulanate: followed of SC and IV cohort without any randomization because the route will be chosen before inclusion by the physician in charge.
  Interventions: Drug: Subcutaneous (SC) route for antibiotic treatment; Drug: Intravenous (IV) route for antibiotic treatment
- ceftriaxone: followed of SC and IV cohort without any randomization because the route will be chosen before inclusion by the physician in charge.
  Interventions: Drug: Subcutaneous (SC) route for antibiotic treatment; Drug: Intravenous (IV) route for antibiotic treatment
- piperacillin-tazobactam: followed of SC and IV cohort without any randomization because the route will be chosen before inclusion by the physician in charge.
  Interventions: Drug: Subcutaneous (SC) route for antibiotic treatment; Drug: Intravenous (IV) route for antibiotic treatment

INTERVENTIONS:
Drug: Subcutaneous (SC) route for antibiotic treatment — Patients receiving one of the three antibiotics by SC route without any randomization because the route will be chosen before inclusion by the physician in charge.
Drug: Intravenous (IV) route for antibiotic treatment — Patients receiving one of the three antibiotics by IV route without any randomization because the route will be chosen before inclusion by the physician in charge.

SUMMARY:
Elderly people are more prone to develop infection with a poorer prognosis compared to young people. Physicians may encounter difficulties regarding antimicrobial agents administration route. In fact, poor venous access and behavioral disturbance are frequent issues. The subcutaneous (SC) route may be a safe alternative, but sparse data are available in the literature. The present study aims to describe Pharmacokinetics (PK) / Pharmacodynamics (PD) characteristics of antibiotics (amoxicillin/clavulanate, ceftriaxone and piperacillin/tazobactam) subcutaneous administration in patients aged over 65.

DETAILED DESCRIPTION:
Antibiotic administration through subcutaneous (SC) injection is common practice in France, especially in Geriatrics as an alternative to intravenous (IV) route in case of poor venous access or delirium (Forestier et al. CMI 2015). Whereas tolerance of such a practice seems to be reasonable (Roubaud-Baudron et al. Age and Ageing 2017), sparse PK/PD data are available. Most PK/PD studies include young and healthy subjects, yet elderly patients often have multimorbidity , poly medication, renal insufficiency and cachexia which may disturb antibiotics PK/PD. Compared to intravenous (IV) route, SC route is less painful and less frequently associated with infectious or thrombotic complication. A recent study carried out in Bordeaux University Hospital comparing PK/PD data on ertapenem SC or IV administrations in patients aged over 75 showed that area under the curve (AUC) and probability to maintain free ertapenem concentration above the Minimum inhibitory concentration (MIC) during at least 40% of time (fT>MIC>40%) were not significantly different (manuscript in progress).

The investigator's hypothesis is that SC administration of amoxicillin-clavulanate, ceftriaxone and piperacillin-tazobactam has favorable pharmacokinetics and acceptable tolerance compared with IV infusion in elderly patients.

Patients receiving one of the three antibiotics by IV or SC route will be included at steady state (depending on antibiotic treatment) for several blood tests (3 or 4 depending of routes choice) and followed until 15 days after completion of antibiotic treatment in order to evaluate tolerance and efficacy of antibiotic treatment. Physicians in charge of patients will decide antibiotic prescription including administration route. The study will not influence these choices because patients will be included after antibiotic initiation.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 65
* To receive ceftriaxone (1g daily) or amoxicillin-clavulanate (1g/0.2g every 8h) or piperacillin-tazobactam (4g/0.5g every 8h) by SC or IV infusion (30-60minutes) at steady state (48h, 24h and 24h respectively)
* Free, written and informed consent signed by the participant or by a proxy in case of delirium

Exclusion Criteria:

* criteria for legislation (justice protection, subject participating to another research including a period of exclusion)
* previous inclusion in this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients will be included during their hospitalization. They may be included if they receive first-line antibiotic treatment or other antibiotic therapy, as long as the time to reach pharmacokinetic steady state has been reached. This project involves patients hospitalized in an infectious and tropical or geriatric ward
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2021-09-05 (Estimated); Study Completion 2021-09-05 (Estimated)

PRIMARY OUTCOMES:
Plasma antibiotic concentrations | Day 1
  Describe and compare pharmacokinetics of amoxicillin-clavulanate, ceftriaxone and piperacillin-tazobactam administered by SC and IV routes

SECONDARY OUTCOMES:
Number of adverse events | Day 21
  Occurrence of adverse events (AEs) up to 15 days after the end of local antibiotherapy (edema, pain, erythema, necrosis) and systemic (AEs described in the Summary of Product Characteristics for antibiotics)
Number of infection cure | Day 21
  rate of infection cure at the end of antibiotic treatment up to 15 days after the end of antibiotic therapy
Number of hospitalisation days | Day 21
  Describe the times of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Claire ROUBAUD-BAUDRON, MD, PhD, Principal Investigator — Hospital University, Bordeaux
Locations (5):
- France (5):
  - CHU de Bordeaux, Bordeaux
  - Hospital Métropole Savoie, Chambéry
  - CHU de Grenoble Alpes, Grenoble
  - Hospices Civils de Lyon, Lyon
  - University Hospital, Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No